CLINICAL TRIAL: NCT04405024
Title: Pilot Study of the Feasibility of Routine Inpatient Hepatitis C Screening
Brief Title: Pilot Study on the Feasibility of Systematic Hepatitis C Screening of Hospitalized Patients
Acronym: HOSPI-VHC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The participating centers were not opened on time, and the inclusion period has expired. A Substantial amendment is in progress to extend the inclusion period.
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Nationale des Hépato-Gastroentérologues des Hôpitaux Généraux (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HOSPI-VHC; 2019-A03309-48 (Other: ID-RCB)
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatitis C testing (Other): If the patient is included in the study, HCV serology (2 x 5 ml tubes) will be taken at the time of admission as part of the routine entry assessment.
  These two tubes will be used for HCV screening. The patient is informed of the HCV serology result during hospitalization by an investigator.
  Interventions: Diagnostic Test: Hepatitis C testing

INTERVENTIONS:
Diagnostic Test: Hepatitis C testing — Hepatitis C Screening

SUMMARY:
The Ministry of Health has set the target of eradicating hepatitis C (HCV) in France by 2025.

The goal is to validate the feasibility and value of conducting routine HCV screening in hospitalized patients.

DETAILED DESCRIPTION:
The number of undetected HCV-infected persons has been extrapolated to 75,000 according to the results of a 2014 study. Screening efforts have been set up in groups of people said to be at high viral risk: drug users, prisoners, precarious persons or migrants from highly endemic countries. Nevertheless, the concept of universal screening has not yet been adopted by the guardians and the Ministry.

It is in this context that "hepatitis free hospital" projects have been carried out in several French cities such as Nice, Nancy and Marseille.

The aim of the HOSPI-VHC study is to evaluate the feasibility and efficiency of systematic HCV screening in all medical and surgical departments of 4 National Association of Hepato-Gastroenterologists of General Hospitals (ANGH) hospitals. This pilot project is part of a public health screening program. It will evaluate the interest and usefulness of implementing universal screening in hospitalized patients without taking into account the existence of viral risk factors. This study will also make it possible to evaluate the implementation of a dedicated care pathway: number of patients screened, number of patients referred for consultation and number of patients accepting the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Hospitalized during the study period
* Non-opposition for participation in the Protocol

Exclusion Criteria:

* Patients under 18 years of age
* Outpatient, long-stay, maternity and intensive care inpatients
* Patients refusing blood collection
* Patient may not understand the information sheet
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2026-06-21 (Estimated)

PRIMARY OUTCOMES:
potential patient versus | 7 days
  Number of HCV serologies collected compared to the number of patients meeting the inclusion criteria during the study period.

SECONDARY OUTCOMES:
HCV positive | 7 days
  Percentage positive for HCV
Follow-up | 2 months
  Percentage of patients referred for consultation if HCV positive
Polymerase chain reaction (PCR) | 7 days
  Percentage of HCV PCR positive patients
Viral risk factor | 7 days
  Percentage of patients with a viral risk factor
hepatic fibrosis | 7 days
  Percentage of patients with hepatic fibrosis
treatment initiation | 2 months
  Percentage of patients benefiting from treatment initiation

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHI Créteil, Créteil
  - Grand Hôpital de l'Est Francilien - Site de Marne-la-Vallée, Jossigny
  - CH Meaux, Meaux
  - CHIV, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No